CLINICAL TRIAL: NCT03380819
Title: Clinical Safety and Efficacy of Pharmacogenetics in Veteran Care
Brief Title: The VetSeq Study: a Pilot Study of Genome Sequencing in Veteran Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Boston Healthcare System (U.S. Federal Agency)
Responsible Party: Principal Investigator, Jason L. Vassy, MD, MPH, SM, Clinician-investigator, VA Boston Healthcare System
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2993
Record Dates: First submitted 2017-12-15; First posted 2017-12-21 (Actual); Last update posted 2023-04-26 (Actual); Status verified 2023-04

CONDITIONS: Rare Diseases; Genetic Disease
MeSH Terms: conditions — Rare Diseases; Genetic Diseases, Inborn

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Genome sequencing (Experimental): Patients undergo exome or whole-genome sequencing, and their patients receive an interpreted clinical report.
  Interventions: Diagnostic Test: Genome sequencing

INTERVENTIONS:
Diagnostic Test: Genome sequencing — Patients will undergo exome or genome sequencing, and their referring provider will receive an interpreted report with the following categories of results: 1) results related to the indication for testing, 2) secondary monogenic results, 3) carrier status, 4) pharmacogenomics results.

SUMMARY:
The VetSeq Study is a pilot intervention study exploring the feasibility of integrating genome sequencing into clinical care at the VA Boston Healthcare System.

DETAILED DESCRIPTION:
The VetSeq Study is a pilot intervention study exploring the feasibility of integrating genome sequencing into clinical care at the VA Boston Healthcare System. Healthcare providers may refer any patients who they think might benefit from diagnostic whole genome or exome sequencing. Providers will briefly discuss genome sequencing and the pilot study with potentially eligible patients. If a patient is interested, the provider will refer him/her to the study by contacting the study staff and providing the reason (clinical question) why the provider thinks genome sequencing might be beneficial for the patient. The study staff will meet with the patient to conduct a baseline interview and survey, obtain informed consent for sequencing, and obtain a blood specimen for sequencing. A clinical laboratory will perform exome or whole-genome sequencing and issue an interpreted genome report including any variant possibly explaining the patient's condition, in addition to secondary monogenic, carrier, and pharmacogenomic results. This report will be sent to the referring provider, who will document the results and associated decision-making in the medical record. Approximately 3 months later, study staff will conduct a follow-up interview and survey with the participating patient.

ELIGIBILITY:
Inclusion criteria:

* Patient referred by provider to study for genome sequencing
* Life expectancy of at least 12 months in the judgment of the referring provider

Exclusion criteria:

* Life expectancy of <12 months
* Inability to give informed consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2017-12-29 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Primary molecular diagnosis | Baseline
  Identification of a genetic variant that explains the patient's indication for sequencing

SECONDARY OUTCOMES:
Secondary genomic results | Baseline
  Pathogenic or likely pathogenic variants in over 4600 genes associated with monogenic disease risk, carrier status variants, and pharmacogenomic results

OTHER OUTCOMES:
Change in clinical management | 3 months
  Evidence that genome sequencing results changed the medical care of the patient
Self-reported health and quality of life | 3 months
  Veterans Rand (VR)-12

CONTACTS AND LOCATIONS:
Overall Officials: Jason L Vassy, MD, MPH, MS, Principal Investigator — VA Boston Healthcare System
Locations (1):
- VA Boston Healthcare System, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
A research data repository will be created from the genome sequence data, genome report data, patient survey data, and data abstracted from medical charts. identified genome sequence data.
Supporting Information: Study Protocol, ICF
Time Frame: Indefinitely
Access Criteria: Interested investigators will obtain institutional review board (IRB)-approval and complete a Combined Data Use-Data Transfer Agreement to access the data repository.